CLINICAL TRIAL: NCT06266728
Title: Performance of Total30 for Astigmatism in Digital Device Users
Brief Title: T30 for Astigmatism in Digital Device Users
Acronym: T30FA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern College of Optometry (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00006733
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-04

CONDITIONS: Contact Lens Complication; Astigmatism; Refractive Errors
Keywords: Total30 for astigmatism; Comfort; Dryness; Visual Analog Scale; Contact Lens
MeSH Terms: conditions — Astigmatism; Refractive Errors

STUDY DESIGN:
Intervention Model Description: This prospective, one-month, three-visit study will refit all participants into TOTAL30 for Astigmatism contact lenses.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Total 30 for astigmatism contact lenses (Experimental): Total30 for Astigmatism Monthly Replacement Contact Lenses
  Interventions: Device: Total30 for Astigmatism Contact Lenses

INTERVENTIONS:
Device: Total30 for Astigmatism Contact Lenses — Participants must be refit into Total30 for Astigmatism Contact Lenses and wear them over the course of this one month study.
  Other Names: Lehfilcon A

SUMMARY:
This study aims to determine if Total30 lenses for astigmatism can be successfully fit in participants who are heavy digital device users.

DETAILED DESCRIPTION:
Extensive computer use is no longer an employment-specific challenge. Use of digital devices in work, home, and leisure settings is now the norm, and it is now socially expected. While the introduction of high-powered computers and digital devices have greatly improved many aspects of modern life, the pervasive use of digital devices has caused some patients to develop a condition known as Digital Eye Strain (DES). DES has been reported to be as high as 93% the population depending upon how the condition is defined, and its severity has been found to increase with increased digital device time. DES is a condition where patients experience symptoms such as glare, accommodative dysfunction, defocus, fatigue, discomfort, and dryness from digital device use, and these dry eye symptoms may also result in decreased quality of life. While dryness symptoms in DES are likely multifactorial (e.g., contact lens use, systemic disease status), much of the dryness symptoms in DES are probably due to tear film evaporation secondary to having a reduced number of blinks per minute while using digital devices.

Contact lens (CL) discomfort affects most CL wearers with discomfort consistently topping the reasons why established CL wearers drop out of CLs. In fact, studies have consistently found that the frequency of CL dropout is around 20% with this dropout frequency staying relatively stable over the past 20 plus years. This static frequency of CL dropout is surprising since there have been a number of dramatic soft CL innovations during this time frame (e.g., widely available daily disposable CLs, silicone hydrogel CL materials with high oxygen transmissibility, new CL surface coatings). CL discomfort and dropout could be affected by significant time spent on digital devices and DES. Maintaining ocular comfort with satisfactory CL performance (comfort, lack of dryness, and overall good vision) is key to overall success. This could be especially important in patients who wear astigmatic CLs, yet the community currently lacks data on this topic.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18- to 40-year-old)
* 0.00 LogMAR visual acuity or better in their habitual CLs or by manifest refraction in both eyes
* Smart phone with text messaging capabilities
* Existing wearers of soft, frequent replacement toric CLs within past 6 months
* Frequent digital device user (e.g., phone, iPad, computer, social media, video streaming, etc.) defined as at least 8 hours of usage per day
* Willing to follow the required wear schedule
* Astigmatism ranging from 0.75 D to 2.50 D in each eye
* Willing to wear their CLs at least 13 hours/day

Exclusion Criteria: Have known systemic health conditions that are thought to alter tear film physiology (e.g., Sjögren's syndrome).

* Have a known history of being diagnosed with dry eye disease
* Have a history of ocular surgery within the past 12 months
* Have a history of severe ocular trauma, active ocular infection or inflammation
* Have a history of viral eye disease
* Currently using isotretinoin-derivatives or ocular medications
* Currently using a dry eye treatment including but not limited to artificial tears
* Currently using rewetting drops daily or occasionally
* If they are pregnant or breast feeding
* Need for spectacle add power of any amount (presbyopic)
* Currently wearing T30fA CLs
* Have a history of wearing hard CLs
* Subjects who show excessive lens oscillation with the T30fA lenses during the fitting process yet show 0.0 logMAR acuity, will be excluded from the study.
* Patients who report unstable vision while wearing their habitual or study CLs (e.g., rotational instability of CLs)
* Willing to not use any artificial tears or dry eye treatments during the study
* Willing to not use rewetting drops during the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-18 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Comfort Scores | Baseline to 1 month of Contact lens wear
  Participants will receive text message surveys on which they will record the comfort of their lenses throughout various points in the day, during different periods of the 1 month study. Scores will be recorded on a scale +/- 50 with +50 being the highest level of comfort and -50 being uncomfortable.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Kannar Eye Care, Pittsburg, Kansas
  - Coldwater VIsion Center, Coldwater, Mississippi